CLINICAL TRIAL: NCT05078229
Title: Efficacy of a Mindfulness-Based Stress Management Program for Allogeneic HCT Caregivers
Brief Title: Evaluating Stress Management Among Allogeneic HCT Caregivers
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCC-20786; R01CA255265 (NIH)
Record Dates: First submitted 2021-09-02; First posted 2021-10-14 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Burden; Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- FOCUS (Experimental): Focusing On mindfulness for Caregivers Under Stress (FOCUS)will consist of six one-on-one, 45-60 minute sessions delivered either in-person (sessions 1-3) or via video conference (sessions 4-6). The first few sessions will primarily focus on how to direct attention to the breath or some object of attention (e.g., parts of the body). As the program progresses, participants are asked to apply these skills to thoughts and emotions. Throughout the treatment, caregivers are reminded to utilize existing coping skills, as well as how to integrate the new skills learned throughout this program for managing stress. Formal mindfulness meditations are conducted within each session, lasting from 7-20 minutes; participants will be asked to practice mindfulness exercises daily.
  Interventions: Behavioral: FOCUS
- Healthy Living (Active Comparator): Healthy Living (HL) will consist of six, 45-60 minute sessions delivered one-on-one; sessions 1-3 in-person on HCT unit and sessions 4-6 via video conference. HL will be based on the American Cancer Society's (ACS) Caregiver Resource Guide.
  Interventions: Behavioral: Healthy Living
- Standard of Care - Enhanced Care (No Intervention): Participants in Enhanced Care will receive treatment consistent with what is offered to all caregivers of allogeneic HCT patients. This entails the option of attending weekly support groups and meeting with social workers as needed. At the baseline session, participants randomized to Enhanced Care will be provided with a modified version of the ACS Caregiver Resource Guide.

INTERVENTIONS:
Behavioral: FOCUS — There will be 6 one on one sessions, either in person or via video conference. The 6 sessions will last between 45-60 minutes. Topics of the sessions will be Mindfulness for the Caregivers, Awareness of Stressors, Skillful Actions, Thoughts, Self-Care and Balance and Planning for the Future. There will be meditation during the sessions and then recommended daily at home mindfulness practice.
  Arms: FOCUS
Behavioral: Healthy Living — There will be 6 one on one sessions, either in person or via video conference. The 6 sessions will last between 45-60 minutes. Topics of sessions will be Overview of Cancer, Eating Well, Exercise, Cancer Prevention, Sleep and Finances.
  Arms: Healthy Living

SUMMARY:
The purpose of the study is to understand whether different stress management interventions impact stress among HCT cancer caregivers and patients.

ELIGIBILITY:
Inclusion Criteria:

* Caregiver Inclusion Criteria:
* Caring for a patient planning to receive an allogeneic HCT at Moffitt
* Intending to remain primary caregiver throughout patient treatment (i.e., will be the caregiver the majority of the time)
* Able to provide informed consent
* Able to read and write in English
* Owns a smartphone and is willing to download the study app
* Patient Inclusion Criteria:
* Receiving an allogeneic HCT at the cancer center
* Able to provide informed consent
* Able to read and write in English

Exclusion Criteria:

* Under 21 years of age
* Unable to provide informed consent
* Unable to read and write in English
* Caregiver is unable to remain primary caregiver throughout patient treatment
* Patient does not receive transplant at Moffitt Cancer Center

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 505 (Estimated)
Dates: Start 2021-09-16 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Caregiver Burden at End of Treatment | Up to 8 Weeks
  Caregiver burden will be measured using the Zarit Burden Interview Short Form (ZBI). The ZBI is 12 items using a 5-point Likert scale assessing caregiver burden. Participants rate burden on a scale of 0 to 4, 0 indicating "rarely" an issue and 4 indicating "nearly always" The ZBI has been validated in populations of cancer caregivers and has demonstrated very good internal consistency and discriminative ability
Caregiver Burden at 2 Month Follow-up | 2 month follow up after end of treatment
  Caregiver burden will be measured using the Zarit Burden Interview Short Form (ZBI). The ZBI is 12 items using a 5-point Likert scale assessing caregiver burden. Participants rate burden on a scale of 0 to 4, 0 indicating "rarely" an issue and 4 indicating "nearly always". The ZBI has been validated in populations of cancer caregivers and has demonstrated very good internal consistency and discriminative ability
Caregiver Burden at 6 Month Follow-up | 6 month follow up after end of treatment
  Caregiver burden will be measured using the Zarit Burden Interview Short Form (ZBI). The ZBI is 12 items using a 5-point Likert scale assessing caregiver burden. Participants rate burden on a scale of 0 to 4, 0 indicating "rarely" an issue and 4 indicating "nearly always". The ZBI has been validated in populations of cancer caregivers and has demonstrated very good internal consistency and discriminative ability
Patient Distress at End of Treatment (CESD) | Up to 8 Weeks
  Patient distress will be measured using the Center for Epidemiological Studies Depression Scale (CESD). The CESD is comprised of 20 4-point Likert scale items and has been commonly used among cancer caregivers. Participants rate how often over the past week they experienced symptoms associated with depression, such as restless sleep, poor appetite, and feeling lonely. Response options range from 0 to 3 for each item (0 = Rarely or None of the Time, 1 = Some or Little of the Time, 2 = Moderately or Much of the time, 3 = Most or Almost All the Time). Scores range from 0 to 60, with high scores indicating greater depressive symptoms.
Patient Distress at End of Treatment (GAD-7) | Up to 8 Weeks
  Patient distress will be measured using the Generalized Anxiety Disorder-7 (GAD-7). The GAD-7 is comprised of 8 items on a 4-point Likert scale and has been used extensively among cancer caregivers. Participants rate the severity of his or her symptoms over the past two weeks. The GAD-7 score is calculated by assigning scores of 0, 1, 2, and 3, to the response categories of "not at all," "several days," "more than half the days," and "nearly every day," respectively, and then adding together the scores for the seven questions
Patient Distress at 2 Month Follow-up (CESD) | 2 Month Follow-up after end of treatment
  Patient distress will be measured using the Center for Epidemiological Studies Depression Scale (CESD). The CESD is comprised of 20 4-point Likert scale items and has been commonly used among cancer caregivers. Participants rate how often over the past week they experienced symptoms associated with depression, such as restless sleep, poor appetite, and feeling lonely. Response options range from 0 to 3 for each item (0 = Rarely or None of the Time, 1 = Some or Little of the Time, 2 = Moderately or Much of the time, 3 = Most or Almost All the Time). Scores range from 0 to 60, with high scores indicating greater depressive symptoms.
Patient Distress at 2 Month Follow-up (GAD-7) | 2 Month Follow-up after end of treatment
  Patient distress will be measured using the Generalized Anxiety Disorder-7 (GAD-7). The GAD-7 is comprised of 8 items on a 4-point Likert scale and has been used extensively among cancer caregivers. Participants rate the severity of his or her symptoms over the past two weeks. The GAD-7 score is calculated by assigning scores of 0, 1, 2, and 3, to the response categories of "not at all," "several days," "more than half the days," and "nearly every day," respectively, and then adding together the scores for the seven questions
Patient Distress at 6 Month Follow-up (CESD) | 6 Month Follow-up after end of treatment
  Patient distress will be measured using the Center for Epidemiological Studies Depression Scale (CESD). The CESD is comprised of 20 4-point Likert scale items and has been commonly used among cancer caregivers. Participants rate how often over the past week they experienced symptoms associated with depression, such as restless sleep, poor appetite, and feeling lonely. Response options range from 0 to 3 for each item (0 = Rarely or None of the Time, 1 = Some or Little of the Time, 2 = Moderately or Much of the time, 3 = Most or Almost All the Time). Scores range from 0 to 60, with high scores indicating greater depressive symptoms.
Patient Distress at 6 Month Follow-up (GAD-7) | 6 Month Follow-up after end of treatment
  Patient distress will be measured using the Generalized Anxiety Disorder-7 (GAD-7). The GAD-7 is comprised of 8 items on a 4-point Likert scale and has been used extensively among cancer caregivers. Participants rate the severity of his or her symptoms over the past two weeks. The GAD-7 score is calculated by assigning scores of 0, 1, 2, and 3, to the response categories of "not at all," "several days," "more than half the days," and "nearly every day," respectively, and then adding together the scores for the seven questions

SECONDARY OUTCOMES:
Patient Healthcare Utilization - Readmissions to the hospital at 6 Month Follow-up | 6 Month Follow-up after end of treatment
  Patient Healthcare Utilization will be measured with readmissions to the hospital
Patient Healthcare Utilization - unexpected clinic visits post discharge at 6 Month Follow-up | 6 Month Follow-up after end of treatment
  Patient Healthcare Utilization will be measured with unexpected clinic visits post discharge

CONTACTS AND LOCATIONS:
Overall Officials: Christine Vinci, PhD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yang MJ, Yepez VV, Brandon KO, Reblin M, Pidala J, Jim HSL, Meyer JS, Gore LR, Khera N, Lau P, Sauls RM, Jones SR, Vinci C. A mindfulness-based stress management program for caregivers of allogeneic hematopoietic stem cell transplant (HCT) patients: Protocol for a randomized controlled trial. PLoS One. 2022 Apr 1;17(4):e0266316. doi: 10.1371/journal.pone.0266316. eCollection 2022. PMID 35363799